CLINICAL TRIAL: NCT04528953
Title: Investigating the Effect of Interval Walking and Qigong on Some Clinical and Biological Outcomes of People With Knee Osteoarthritis.
Brief Title: Investigating the Effect of Interval Walking and Qigong on People With Knee Osteoarthritis: Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00146006
Record Dates: First submitted 2020-08-11; First posted 2020-08-27 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interval group (Experimental)
  Interventions: Behavioral: Interval walking and Qigong exercise
- Qigong exercise (Experimental)
  Interventions: Behavioral: Interval walking and Qigong exercise
- continuous walking (Active Comparator)
  Interventions: Behavioral: Interval walking and Qigong exercise

INTERVENTIONS:
Behavioral: Interval walking and Qigong exercise — Interval walking: The subjects will be asked to complete daily 30 minutes of walking in two 15-minute bouts with the rest interval for at least 0.5 an hour and not more than 2 hours between each bout.
  Qigong exercise: mind-body exercise using the "six healing sound" Qigong exercise will be used because it is easy to learn, requires minimal physical capability, and can be performed even in a sitting body position.

SUMMARY:
Knee osteoarthritis (KOA) causes pain and limited function that leads to a sedentary lifestyle. The sedentary lifestyle increases the risk of cardiovascular diseases. In addition, many subjects with KOA have knee pain and sleep disturbance that limit their function, quality of life and cause body fatigue. Walking exercise can benefit people with KOA. However, continues walking for more than 30 minutes can increase pain that may stop people from participation in walking exercise.

Interval walking may complete the same amount of walking exercise in several separate time periods, without causing extra pain in people with KOA. Mind-body exercise may improve sleep and pain in people with KOA.

This study will help researchers to find out whether the interval walking, or mind-body exercise may help people with KOA to improve their pain, fitness level, sleep quality, exercise participation, fatigue, and quality of life.

By doing this study, researchers hope to learn more about the interval walking or mind-body exercise in people with KOA.

ELIGIBILITY:
Inclusion criteria are the following:

1. 60-79 years of age and diagnosed with KOA by a physician or meet the ACR criteria (95% sensitivity, and 69% specificity) for KOA. The ACR criteria include experiencing almost daily knee pain and having at least 3 of these 6 criteria: (1) Age more than 50 years old, (2) less than 30 minutes of morning stiffness, (3) increased warmth of the knee, (4) crepitus with flexion or extension, (5) joints' bony enlargement , and (6) tenderness of joint line with palpation, or subject must be diagnosed radiologically, with grade II or more according to the Kellgren and Lawrence rating scale.
2. Frequent knee pain or aching on most of the preceding 30 days.
3. An average of mild to moderate pain intensity level (5 to 75 mm on the 100 mm VAS) in the last 7 days
4. Sedentary lifestyle assessed using 2011 Compendium of Physical Activities questionnaire. The subject is considered sedentary if engaging in exercise or physical activity with metabolic equivalents of task (MET) less than 4, not more than two times/week.

Exclusion criteria:

1. Unwilling to attend 3 sessions/week at Kirmayer Fitness Center
2. Having other types of arthritis such as rheumatoid arthritis or gout
3. Neurological disorders
4. CVD including hypertension that prevent them from engaging in walking exercise
5. Currently using beta blocker medication
6. Underwent any lower limb surgery during the past 6 months
7. A history of two or more incidents of fall during the last 6 months
8. Current hip or spine pain that prevents them from engaging in walking exercise.

Ages: 45 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility measurement: recruitment, compliance, and dropout | 6 week
  Feasibility will be quantified using rates of participant recruitment, compliance, and dropout rate from the exercise program using exercise diary filled by the exercise supervisor. The Percentage of recruited subjects per month will be reported. The dropout rate is defined as the percentage of subjects who do not complete the study intervention and choose to withdraw. The compliance is defined as the percentage of the completed exercise program. The exercise diary log of subjects who drop out of the study will not be included when compliance is calculated. (feasibility measures will be reported in percentage)
Acceptability | 6 week
  Acceptability will be assessed via participants' program evaluation scores and rating of treatment satisfaction at the end-intervention evaluation. The subjects will be asked to score, on an 11-point scale, ranging from 0 (poor) to 10 (excellent) for questions "How do you rate this exercise program overall in regarding to ease of use?" and "How do you rate this exercise program overall in regarding to improving your symptoms?" Participants will be also asked to rate their overall level of satisfaction with the intervention using an 11-point numerical rating scale ranging from 0 (completely dissatisfied) to 10 (completely satisfied).

SECONDARY OUTCOMES:
Comprehensive pain assessment: the Measure of Intermittent and Constant Osteoarthritis Pain | 6 week
  For comprehensive pain assessment: The Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP) scale. ICOAP is a multidimensional measure developed to evaluate the pain in subjects with KOA, comprehensively. ICOAP assesses both pain intensity and frequency in addition to assessing the impact of pain on sleep, and quality of life (physical function). ICOAP has high reliability (0.85) and validity (0.60-0.81). ICOAP is 11-points scale to assess OA pain with maximum score 100.
Resting heart rate (rHR) and heart rate recovery (HRR) | 6 week
  rHR and HRR will be measured using a Polar OH1 optical HR sensor (Polar Electro Inc., New York), which is in high agreement with ECG measured HR and is validated to be used in lab sittings. HRR is defined as the range of the change of HR from the peak after the exercise to one-minute post-exercise. Slow HRR is a warning of decline of cardiovascular/autonomic function. The HR should decrease at least 12 beats after one minute after exercise termination, otherwise this is considered as an abnormal response. The HRR will be measured post the 6-minute walk test, which has been approved to be as effective in testing HRR as vigorous exercises. The HR will be measured before the exercise (rHR), immediately after the exercise (the peak HR), and one minute after the exercise(1-min-post). Then, the difference between the peak HR and the 1-min-post will be calculated.
Heart rate variability (HRV) | 6 week
  HRV will be estimated using an ECG system via analyzing the HRV frequency and time domain. Standard lead II configuration will be used by placing three disposable electrodes over the participant's chest to record the ECG signals. We will collect the ECG signal at 2000 Hz sampling rate.The subject will be asked to sit relaxed in a quiet room with a temperature between 22 and 24°C, for 10 minutes. Then, the HRV ECG recording will be collected over a 5-minute period while participants are asked to not move or speak over the next 5 minutes when HRV will be collected. BIOPAC AcqKnowledge 5.0 software will be utilized to collect both the frequency and the time parameters of HRV. The frequency parameters are LF power (0.04-0.15 Hz) and HF power (0.15-0.4 Hz) and LF/HF ratio, while the time parameters includes RMSSD.
Blood pressure | 6 week
  SBP will be measures using an automatic device, Microlife BP monitor.
insomnia severity | 6 week
  Insomnia Severity Index is a 7-item questionnaire that is a global measure of perceived insomnia severity, with its reliability and validity have been reported.
Sleeping Quality: Pittsburgh Sleep Quality Index | 6 week
  Sleeping Quality Assessment will use Pittsburgh Sleep Quality Index (PSQI) with high test-retest reliability and construct validity.
Fatigue: Multidimensional Fatigue Inventory (MFI-20) | 6 week
  Fatigue will be measured using Multidimensional Fatigue Inventory (MFI-20), with proved internal consistency, validity, and utilized in research of OA.
Depression: Geriatric Depression Scale | 6 week
  The 15-item questionnaire of the Geriatric Depression Scale will be used, which is a valid measurement of depression.
Knee Injury and Osteoarthritis Outcome Score | 6 week
  Injury and Osteoarthritis Outcome Score (KOOS) is a valid and reliable instrument and will be used for short-term and long-term follow-up of knee OA. KOOS consists of 42 items. A Likert scale is used for each sub-scale and items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale. Zero representing extreme knee problems and 100 representing no knee problems.
  in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
36 short form Quality of Life | 6 week
  The SF-36 measures eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Inflammatory biomarkers | 6 week
  The inflammatory biomarker assessments will use venous blood samples drawn from subjects. Approximately 10 ml of blood will be collected from fasting subjects, between 8 am to 10 am. The serum will be assayed for the levels of inflammatory markers: TNF-α, IL-1β, IL-6, IL-8, IL-17, and C-reactive protein, using respective ELISA kits available from Thermo Scientific, Inc (Rockford, IL).
Fitness level- The 6-minute walk test | 6 week
  The 6-minute walk test will be used to assess the fitness level at the baseline and after completing the intervention. We will follow the guideline of the American Thoracic Society to conduct this test as the improvement in walking distance indicates the improvement of aerobic fitness.
Pain intensity measurement | 6-week
  Pain intensity level will be assessed using 100 mm horizontal VAS, which is a valid and reliable pain scale. The VAS is reported to be a sensitive measurement to hourly and weekly assessment of pain level, and a reduction of 10mm is reported to be the minimum clinical important difference for people with chronic pain such as in OA. The subjects in both groups will be asked to score their pain before and after each session of the walking exercise, and the averaged range of change from pre to post walking will be used in data analysis.
  In addition, for change of pain from baseline to post intervention, the participant will be asked to report their minimum and maximum pain during the last 24 hours, and their current pain on the VAS ruler. Then, the average of the measure taken 3 different times will be used in the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Wen Liu, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No